CLINICAL TRIAL: NCT07264595
Title: A Study to Evaluate the Safety and Tolerability of Multiple Ascending Doses of GS3-007a Dry Suspension in Patients With PGHD and to Evaluate the Efficacy and Safety of 52-week of Treatment With GS3-007a Dry Suspension: a Two-part, Multicenter, Randomized, Phase Ib/II Clinical Trial
Brief Title: A Study (Phase 1b/2) of GS3-007a Oral Treatment in Children With Growth Hormone Deficiency (PGHD)
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: GenSci073-201
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Pediatric Growth Hormone Deficiency
Keywords: GS3-007a dry suspension; PGHD

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose Level 1~ Dose Level 4 (Placebo Comparator): dose level 1、dose level 2、dose level 3、dose level 4
  Interventions: Drug: GS3-007a dry suspension; Drug: Placebo for GS3-007a dry suspension
- Cohort 1~ Cohort 3 (Active Comparator): GS3-007a low dose , GS3-007a high dose , rhGH 0.033mg/kg
  Interventions: Drug: GS3-007a dry suspension; Drug: rhGH injection
- GS3-007a cohort (Experimental): GS3-007a optimal dose
  Interventions: Drug: GS3-007a dry suspension

INTERVENTIONS:
Drug: GS3-007a dry suspension — GS3-007a
  Other Names: GS3-007a
Drug: Placebo for GS3-007a dry suspension — Placebo for GS3-007a dry suspension
  Other Names: placebo
  Arms: Dose Level 1~ Dose Level 4
Drug: rhGH injection — rhGH injection
  Other Names: rhGH
  Arms: Cohort 1~ Cohort 3

SUMMARY:
This is a two-part clinical study for children with growth hormone deficiency. In the first part, participants will be randomly assigned to receive different doses of an oral treatment (GS3-007a dry suspension) or a placebo for 14 days. This part is double-blinded, meaning neither the participants nor the doctors will know who is receiving the treatment or placebo. The goal is to find a safe and well-tolerated dose.

In the second part, participants will be randomly assigned to receive either the selected dose of GS3-007a or another approved treatment for 52 weeks. This part is open-label, so everyone will know which treatment is being given. After that, all participants may continue taking GS3-007a for another 156 weeks in an extension phase to study long-term effects.

ELIGIBILITY:
Inclusion Criteria:

* chronological age (CA) ≥3 years at Screening
* Prepubertal girls or boys
* Height at Screening lower than the reference height for normal children of the same chronological age and sex minus 2 standard deviations (-2 SD)
* A confirmed diagnosis of growth hormone deficiency (GHD)
* Having not been treated with any growth-promoting drugs
* BA delayed by ≥6 months compared with the CA at Screening Subjects who meet all of the following criteria are eligible to enroll in the extension study (applicable for Part II extension period)
* Subjects who have completed the 52-week treatment period of phase II
* Subjects who do not permanently discontinue the investigational Medicinal Product (IMP) during the 52-week treatment period of phase II

Exclusion Criteria:

* A highly allergic constitution
* Suspected or confirmed total pituitary deficiency, including patients previously confirmed with deficiency of ≥2 pituitary hormones other than GH
* Being confirmed with other chromosomal abnormalities or growth abnormalities affecting growth
* Congenital skeletal dysplasia or serious spinal anomalies
* Cognitive hypofunction, neurodevelopmental disorders, or psychiatric/psychological disorders that, in the investigator's opinion, may interfere with evaluation of study endpoints
* Any clinically significant abnormality that may affect growth or evaluation of the IMP
* Screening magnetic resonance imaging (MRI) scan of the sellar region confirming prior or current intracranial tumor growth
* Concurrent use of any medications that may affect growth or response to growth hormone therapy
* Epiphyseal closure
* Electrocardiogram (ECG) QTcF interval abnormal, with a history of QT/QTc interval prolonged
* Hepatic function indicators abnormal at Screening Patients meeting any of the following criteria may not be enrolled in this extension study (applicable for Part II extension period)
* Subjects with closed epiphyses
* Any clinically significant abnormality that may affect growth or evaluation of the IMP
* Known or suspected allergy to the IMP
* Women with positive blood human chorionic gonadotropin (hCG) at the pre-treatment visit

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2030-11 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events (TEAEs) | up to 21 days (Ib phase)
Annualized height velocity (AHV) at Week 26 of treatment | 26 weeks (II phase)
Number of Participants With TEAEs | up to 160 weeks (II phase extension)

SECONDARY OUTCOMES:
PK concentrations of GS3-007a and metabolite GS3-017 | up to 7 days (Ib phase)
Concentrations of serum growth hormone (GH), insulin-like growth factor-1 (IGF-1), and insulin-like growth factor-binding protein 3 (IGFBP-3) | up to 14 days (Ib phase)
AHVs at each evaluation point | 13 weeks, 39 weeks, 52 weeks (II phase)
Changes from baseline (ΔIGF-1 SDS) in the standard deviation score of the PD indicator insulin-like growth factor-1 (IGF-1 SDS) at each evaluation point | 4 weeks, 13 weeks, 26 weeks, 39 weeks, 52 weeks (II phase)
AHVs at each evaluation point | up to 156 weeks (II phase extension)
Change from extension baseline in the height standard deviation score at each evaluation point (ΔHT SDS) | up to 156 weeks (II phase extension)

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei, China